CLINICAL TRIAL: NCT03033550
Title: A Single-arm Proof of Concept, Open Trial Clinical Study Investigating the Feasibility and Efficacy of Integrating Behavioral and Mobile Health Educational Interventions for Primary and Secondary Prevention in the Primary Care Setting
Brief Title: Integrating Primary & Secondary Interventions for Cervical Cancer Prevention in Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Natalie Pierre-Joseph, Assistant Professor of Pediatrics, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-34457
Record Dates: First submitted 2017-01-13; First posted 2017-01-27 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: HPV-Related Carcinoma
Keywords: HPV vaccination; Cervical cancer screening; Primary care setting; Primary prevention of cervical cancer; Secondary prevention of cervical cancer; Mobile health information

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single (Experimental): single arm- behavioral educational intervention of a brief negotiated mobile application
  Interventions: Behavioral: brief negotiated mobile application

INTERVENTIONS:
Behavioral: brief negotiated mobile application — The intervention will supplement the standard of care with the following steps: (1) mobile- based brief negotiated Intervention ( BNI); (2) a customized companion communication vaccine report to be given before AFG sees provider; and (3) automated interactive Electronic Recall/Reminder Messages (Text messaging), including text messaging and access to a website which includes information about HPV, HPV Vaccine, and cervical cancer screening guideline.

SUMMARY:
The purpose of this study is to determine whether a mobile health educational intervention for Human PapillomaVirus (HPV) Vaccination promotion and cervical cancer screening in Primary Care settings is a feasible behavioral intervention to integrate as a primary and secondary cervical cancer prevention approach.Study Design: The investigators will conduct an open feasibility proof-of-concept trial using a single experimental group with all subjects receiving the behavioral intervention being studied.

Outcome measures. The primary outcome of interest is receipt of the first dose and completion of the three-dose series of HPV vaccine within 6 month of intervention, this will be evaluated by Electronic medical review review.

DETAILED DESCRIPTION:
Background: Nearly 80 million people in the US are infected with HPV and 14 million new cases are diagnosed annually. There is an increasing HPV prevalence among women through the young adult years. Although the body clears many HPV infections persistent infections can progress to cancer and other HPV-related diseases. Cervical cancer is the most common cancer caused by HPV.

Many of the HPV-associated cancers are preventable with a series of safe and effective HPV vaccines. To date, no state has attained the 80% target vaccination rate for HPV. Despite the proven benefits and safety of HPV vaccine, usage remains suboptimal (only 38% had completed the three-dose series) and lower than other recommended adolescent vaccines.

Objective/Hypothesis: Our short term objective is to increase HPV vaccine initiation and completion rates among all age-eligible adolescent girls for whom vaccine is not contraindicated; and explore and examine acceptability of providing HPV vaccination to female youth during her adult female guardian's (AFG) cervical cancer screening appointment.

The investigators hypothesize that a combined intervention which includes (1) a motivational web-based education aimed at AFGs and youth females in their Primary Care site; and (2) text message reminders and an informational web-link on HPV vaccine and cervical cancer screening will increase HPV vaccination rates among youth females and will increase cervical cancer screening rates among their respective AFGs.

The investigators propose the following Aim:

Specific Aim: Conduct a single-arm proof of concept, open trial clinical study investigating the feasibility and efficacy of integrating primary and secondary prevention model for HPV and cervical cancer: a mobile educational and automated electronic interactive messaging intervention that will remind AFG and youth females of scheduled and missed second and third HPV vaccination appointments, and deliver brief text and video educational messaging on HPV, HPV vaccine, and cervical cancer screening.

Study Design: The investigators will conduct an open feasibility proof-of-concept trial using a single experimental group with all subjects receiving the behavioral intervention being studied.

Outcome measures. The primary outcome of interest is receipt of the first dose and completion of the three-dose series of HPV vaccine within 6 month of intervention, this will be evaluated by Electronic medical review review.

ELIGIBILITY:
Inclusion Criteria:

* AFG ages 30 years and older who receive primary care at the study sites.
* AFG consent to have cervical cancer screening status checked in Electronic Medical Record.
* AFG has a daughter between the ages of 11 to 17 who receive primary care at either
* Family Medicine or Pediatric and Adolescent primary care clinic at Boston Medical Center.
* AFG consent to have daughter's HPV vaccination status checked in Electronic Medical Record.
* AFG's daughter has neither initiated the HPV vaccine nor completed the three vaccine series
* AFG and daughter have the ability to read and write in English.
* AFG and daughter each have a cell phone with text messages capabilities.

Exclusion Criteria:

* The investigators will exclude based on the following criteria:
* AFG being seen for a sick visit.
* AFG has an adolescent daughter who is pregnant or is a mother.
* AFG has a daughter who has completed the three dose HPV vaccine series.
* AFG, in the opinion of the clinical staff, is cognitively impaired and unable to give informed consent and may not participate.

Ages: 9 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Number of participants who received the first dose and completed the vaccine series as measured electronic medical record review | up to 6 months
  The primary outcome of interest is receipt of the first dose and completion of the three or two-dose series of HPV vaccine by participants within 6 month of intervention, this will be evaluated by Electronic Measure Review. Unit of measure: Number of participants who received the first doses and who competed the total number of does based - recorded as percentage who receive the first dose, and completed the two or 3 doses.

SECONDARY OUTCOMES:
Patient knowledge and provider-patient communication | over 6 months
  The secondary outcomes are: (a) Change in knowledge of HPV, HPV vaccination, and cervical cancer screening as evaluated by pre/post intervention survey: unit of Measure: based on a 1-10 point scale, with 10 being the highest score;
provider communication about HPV vaccine | through study completion, an average of 1 year
  greater provider communication about HPV vaccine : Unit of measure- the number of participants who responded yes to provider communication about HPV vaccine

OTHER OUTCOMES:
Cervical cancer screening rate | through study completion, an average of 1 year
  Cervical cancer screening rate as evaluated by Electronic Medical Review review: Unit of Measure: Number of participants who has cervical cancer screening within the time guideline ( as measured and reported as percentage who screened within the pap smear guideline

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Joseph, MD MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No